CLINICAL TRIAL: NCT03834714
Title: Effects of Noise Exposure and Near Infrared Light (NIL) on Auditory Health and Performance
Brief Title: Noise Exposure and Near-Infrared Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Office of Naval Research (ONR) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael E. Hoffer, Professor, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 20181214; GR014085 (Other Grant/Funding Number: Office of Naval Research)
Record Dates: First submitted 2019-02-05; First posted 2019-02-08 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Hearing Loss, Noise-Induced
Keywords: Noise induced hearing loss; Near infrared energy; Hering test
MeSH Terms: conditions — Hearing Loss, Noise-Induced

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Noise Stimulus and Infrared Light (Active Comparator): All participants will receive noise stimulus at each of the 4 visits. In addition, they will receive infrared light therapy for 2 out of the 4 visits and sham infrared light therapy for the other 2 visits.
  Interventions: Device: Near Infrared Light; Other: Noise Stimulus
- Noise Stimulus and Sham (Sham Comparator): All participants will receive noise stimulus at each of the 4 visits. In addition, they will receive sham infrared light therapy for 2 out of the 4 visits and infrared light therapy for the other 2 visits.
  Interventions: Other: Noise Stimulus; Device: Sham Near Infrared Light

INTERVENTIONS:
Device: Near Infrared Light — NIR Light Therapy will be administered with the Earlight Generation 1.4 device during 2 out of the 4 sessions. It will be administered to each ear individually for 30 minutes per ear.
  Arms: Noise Stimulus and Infrared Light
Other: Noise Stimulus — Noise stimulus will be administered, open ear, to continuous broadband noise up to 25% of the allowable daily dose of noise per the AFI 48-127 Occupational Noise and Hearing Conservation Program.
Device: Sham Near Infrared Light — Sham NIR Light Therapy will be administered with the Earlight Generation 1.4 device during 2 out of the 4 sessions. It will be administered to each ear individually for 30 minutes per ear.
  Arms: Noise Stimulus and Sham

SUMMARY:
The primary objective of this work is to determine the effect noise has on the auditory system (both auditory health and performance) and also the degree to which the effect of pre-noise therapy such as Near Infrared (NIR) light can mitigate the effects of noise exposure.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old, male or female
* Pass hearing exam with a threshold of 25 decibels (dB) hearing or less, for each ear, for all frequencies tested from 500 Hz to 8000 Hz
* Normal otoscopic exam, otoacoustic emissions (OAEs), and middle ear function as demonstrated by a normal tympanogram
* Completion of a hearing history questionnaire

Exclusion Criteria:

* Screening hearing test failure
* Pregnant females
* Adults unable to provide consent
* History of significant ear surgery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Change in auditory threshold | Baseline, up to 365 days
  Auditory function tests will be measured through the change in air conduction threshold measurements from 500 up to 8000 Hz

SECONDARY OUTCOMES:
Change in otoacoustic emissions (OAE) | Baseline, up to 365 days
  Auditory performance will be measured through OAE testing
Change in central auditory performance (CAP) | Baseline, up to 365 days
  Auditory performance will be measured through central auditory processing assessments

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Hoffer, MD, Principal Investigator — University of Miami
Locations (3):
- United States (3):
  - U.S. Army Aeromedical Research Laboratory, Fort Rucker, Alabama
  - University of Miami Miller School of Medicine, Miami, Florida
  - Wright-Patterson Air Force Base, Wright-Patterson Air Force Base, Ohio

IPD SHARING:
Plan to Share IPD: No